CLINICAL TRIAL: NCT04553562
Title: Efficacy of Acupuncture for Female With Non-cyclic Chronic Pelvic Pain: a Three-armed Randomized Controlled Trial
Brief Title: Acupuncture for Female With Non-cyclic Chronic Pelvic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Principle investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-248-KY
Record Dates: First submitted 2020-09-06; First posted 2020-09-17 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Chronic Pelvic Pain
Keywords: Acupuncture; Sham acupuncture; Randomized controlled trial; Non-cyclic chronic pelvic pain
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants in the acupuncture and sham acupuncture will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture group (Experimental): For acupuncture group, sterile adhesive pads will be placed after skin disinfection on the acupoints. Guanyuan (CV4)，Qihai (CV6)，bilateral Sanyinjiao (SP6), Yinbao (LR9), Qixue (KI13) and Fujie (SP14) will be inserted through the pads. The participants will be treated three times a week, on alternate days, for 6 successive weeks; 18 sessions for each patient in total.
  Interventions: Device: Acupuncture
- Sham acupuncture group (Sham Comparator): For the sham acupuncture group, aterile adhesive pads will be placed after skin disinfection on the acupoints and needles with a blunt tip will be inserted at the same acupoints in the acupuncture group without penetrating the skin.No manipulation of needles will be conducted. The participants will be treated three times a week, on alternate days (ideally), for 6 successive weeks; 18 sessions for each patient in total.
  Interventions: Device: Sham acupuncture
- Waiting list group (No Intervention): For the waiting list group, patients will receive no treatment in the first 6 weeks and will receive the same treatment used in the acupuncture group according to patients' preference.

INTERVENTIONS:
Device: Acupuncture — Sterile adhesive pads will be placed after skin disinfection on the acupoints. Guanyuan (CV4)，Qihai (CV6)，bilateral Sanyinjiao (SP6), Yinbao (LR9), Qixue (KI13) and Fujie (SP14) will be inserted through the pads by the needles (0.30mm in diameter, 40 mm in length, Hwato Brand, Suzhou Medical Appliance Factory, China) to a depth of 25-30mm. Yintang (GV4) will be inserted through the pads by the needle (0.30mm in diameter, 25mm in length, Hwato Brand, Suzhou Medical Appliance Factory, China) to a depth of 10-15mm. The needles at all points will be lightly lifting, thrusting, and twirling every 10 minutes during each session with the sensation of sourness, achiness, heaviness and numbness (deqi). The participants will be treated three times a week, on alternate days (ideally), for 6 successive weeks; 18 sessions for each patient in total.
  Arms: Acupuncture group
Device: Sham acupuncture — Sterile adhesive pads will be placed after skin disinfection on the acupoints. Needles (0.30 mm in diameter, 25 mm in length) with a blunt tip will be inserted at the Guanyuan (CV4)，Qihai (CV6)，bilateral Sanyinjiao (SP6), Yinbao (LR9), Qixue (KI13) and Fujie (SP14) without penetrating the skin. The participants will be treated three times a week, on alternate days (ideally), for 6 successive weeks; 18 sessions for each patient in total.
  Arms: Sham acupuncture group

SUMMARY:
Chronic pelvic pain (CPP) is one of the common symptoms of women at childbearing age. The aim of this study is to assess the efficacy of acupuncture for female with non-cyclic chronic pelvic pain. A three-arm randomized controlled trial (RCT) using acupuncture, sham acupuncture and waiting list with a total sample of 150 will be conducted.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is a persistent pain in pelvis, anterior abdominal wall, lower back, or buttocks lasting at least six months. According to a WHO epidemiological study, the worldwide prevalence rate of CPP in childbearing age women was 2.1%-24%. At present, nearly 55% of the patients had unclear etiology, and there is no universally accepted diagnosis, evaluation and treatment. CPP is often associated with gynecological and non gynecological diseases, including endometriosis, abdominal visceral adhesion, myofascial pain and dysfunction, irritable bowel syndrome and interstitial cystitis/bladder pain syndrome. CPP are also accompanied by psychological and physiological dysfunction, the most common is depression and anxiety, which seriously affects the quality of life of patients.

Acupuncture may have effect on non-cyclic CPP in female, however, there is a lack of evidence of effectiveness of acupuncture. A multi-center randomized three-armed controlled trial will be conducted. The aim of this study is assess the efficacy and safety of acupuncture for female patients with non-cyclic CPP.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of non-cyclic CPP.
* Age 18 to 50 years.
* Have moderate to severe pain in pelvis, anterior abdominal wall, lower back, or buttocks lasting at least six months.
* The mean degree of pelvic pain in the past week rated by Visual Analogue Scale is ≥40 scores.
* Sign informed consent and participate in the study voluntarily.

Exclusion Criteria:

* Have endometriosis (including adenomyosis), ovarian cyst (larger than 3cm), hysteromyoma (larger than 3cm), severe pelvic adhesion, pelvic malignant tumor (relevant examination must be within the last 6 months).
* Have acute pelvic/urinary tract infection.
* Have pain after pelvic surgery.
* Have recurrent gastrointestinal or bladder diseases such as irritable bowel syndrome, interstitial cystitis / bladder pain syndrome, etc.
* During pregnancy or in lactation or have a pregnancy plan within 8 months.
* Have heart, lung, liver, kidney, mental disorders or cognitive dysfunction.
* Have acupuncture treatment in recent 3 months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The change from baseline of the mean score in the past week of the Visual Analogue Scale | Week 6, 18 and 30
  The scores of the Visual Analogue Scale range from 0 to 10，higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The change from baseline of the Brief Pain Inventory score | Week 6, 18 and 30
  The Brief Pain Inventory score uses 0-10 numeric scales for item rating with 0 being "no pain" and 10 being "pain as bad as you can imagine". The pain severity score is calculated from the four items about pain intensity with a range from 0 to 40. The pain interference score corresponds to the item on pain interference with a range from 0 to 70. Higher scores of the Brief Pain Inventory mean a worse outcome.
The change from baseline of the pain severity score of the Brief Pain Inventory | Week 6, 18 and 30
  The pain severity score of the Brief Pain Inventory is calculated from the four items about pain intensity. Each item is rated from "no pain" to "pain as bad as you can imagine", and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score corresponds to the item on pain interference. Higher scores of the The pain severity score mean a worse outcome.
The change from baseline of the pain interference score of the Brief Pain Inventory | Week 6, 18 and 30
  The pain interference score of the Brief Pain Inventory corresponds to the item on pain interference. The seven subitems are rated from "does not interfere" to "completely interferes", and contributes with the same weight to the final score, ranging from 0 to 70. Higher scores of the pain interference score mean a worse outcome.
The proportion of patients with decrease of 0.6 score or more from baseline of the pain interference score of the Brief Pain Inventory | Week 6, 18 and 30
  The pain interference score of the Brief Pain Inventory corresponds to the item on pain interference. The seven subitems are rated from "does not interfere" to "completely interferes", and contributes with the same weight to the final score, ranging from 0 to 70. Higher scores of the pain interference score mean a worse outcome.
The proportion of patients with decrease of 20% or more from baseline of the pain severity score of the Brief Pain Inventory | Week 6, 18 and 30
  The pain severity score of the Brief Pain Inventory is calculated from the four items about pain intensity. Each item is rated from "no pain" to "pain as bad as you can imagine", and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score corresponds to the item on pain interference. Higher scores of the The pain severity score mean a worse outcome.
The change from baseline of the Pain Catastrophising Questionnaire score | Week 6, 18 and 30
  The Pain Catastrophising Questionnaire is a validated scale with 13 items, each scored from 0 (not at all) to 4 (all the time) with a total score range of 0-52, across three domains: rumination (0-16); magnifications (0-12); and helplessness (0-24).Higher scores of the Pain Catastrophising Questionnaire mean a worse outcome.
The change from baseline of the Hospital Anxiety and Depression Scale score | Week 6, 18 and 30
  the score of the Hospital Anxiety and Depression Scale ranges from 0 to 42. Higher scores mean a worse outcome.
The change from baseline of the World Health Organisation Quality of life - Bref Questionnaire score | Week 6, 18 and 30
  Domain scores for the World Health Organisation Quality of life-Bref Questionnaire score are calculated by taking the mean of all items included in each domain and multiplying by a factor of four. These scores are then transformed to a 0-100 scale.Higher scores denote higher quality of life.
The proportions of participants in each response category of the Patient global impression of change | Week 6, 18 and 30
  Patient global impression of change consists of 7 response categories with a range of 1-7: "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." Higher scores mean a worse outcome.
The proportion of subjects using rescue medications and the duration of medication use | Week 6, 18 and 30
  The use of medications during this trial. However, medication use is allowed for intolerable symptoms as long as it is recorded accordingly, including the name, the dosage, and the duration of the medication use.

OTHER OUTCOMES:
Blinding assessment | Week 6
  To test the success of blinding, participants in the acupuncture group and the SA group will be asked to reply to the following question at the 6th week of treatment (sessions 18): "Do you think you have received traditional acupuncture in the past weeks?" The participants will be able to choose one of the following options as the answer: "Yes", "No" or "Unclear".
Safety assessment | Week 0 to 30
  We will handle and document the adverse events (AEs) using the standard operating procedures for monitoring and reporting all AEs. According to their potential association with the treatment, AEs will be categorized as treatment-related or non-treatment-related within 24 hours after their occurrence. Treatment-related AEs include pain, haematoma, localized infection, broken needle, fainting, nausea, headache, dizziness, insomnia, vomiting, or palpitations during or after treatment. In addition, adverse events that are irrelevant to the treatment will be recorded during the study period.
Expectation of improvement assessment | Baseline
  Patients choosing "improved" in the expectation assessment will be asked: "To what extent do you think your pelvic pain will be helped after acupuncture treatment?" Participants will choose the answer from the following options: a great degree, a moderate degree, a small degree, unclear.
Trust evaluation of acupuncture therapy | Baseline and week 6
  Patients choosing "improved" in the expectation assessment will be asked: "To what extent do you think your pelvic pain will be helped after acupuncture treatment?" Participants will choose the answer from the following options: a great degree, a moderate degree, a small degree, unclear.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, PhD, Study Chair — Guang'an men hospital, China Academy of Chinese Medical Sciences